CLINICAL TRIAL: NCT02323750
Title: Systolic Dysfunction to Congestive Heart Failure Cohort Study
Brief Title: TransitionCHF Systolic Dysfunction to Congestive Heart Failure Cohort Study
Acronym: TransitionCHF
Status: Active, not recruiting | Type: Observational
Sponsor: University of Göttingen (Other)
Collaborators: University Medical Center Goettingen (Other); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Gerd Hasenfus, Prof. Dr. med. Gerd Hasenfuß, University of Göttingen
Other Study IDs: TransitionCHF
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Systolic Dysfunction, Transition, Heart Failure, Biobank
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Up to 100 mL blood and 40 mL urine are received for each patient at baseline and one follow-up. Samples are managed through the DZHK Heart bank collection (https://dzhk.de/en/dzhk-heart-bank).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
TransitionCHF aims to recruit a unique cohort of patients with asymptomatic left ventricular dysfunction (NYHA I) to study the progression to symptomatic (>NYHA I) HF and to identify parameters/ biomarkers promoting and predicting the individual risk of transition. Results from TransitionCHF Cohort Study will inform and refine current treatment guidelines. The implementation of common patient data sets and biobanking standards will enable data and biomaterial sharing with other study groups of the German Center for Cardiovascular Research (DZHK). This study will set the standard for a unique DZHK heart failure database and Biobank for innovative preclinical and clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic systolic dysfunction (defined as: ejection fraction < 40% by echocardiography or MRI; documented within the last 3 months prior to baseline visit)
* A maximum of one hospitalization for heart failure (defined as hospitalization with signs and symptoms of heart failure requiring intravenous loop diuretic therapy within 48 hours after hospital admission) at least 2 years prior to the baseline visit
* No heart failure symptoms (NYHA II, III or IV) upon inclusion
* 6MWD ≥ 80% of reference values
* Written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Symptomatic heart failure (NYHA>I) at baseline visit
* Any significant valvular disease (> 2nd degree)
* Severe pulmonary disease (e.g. FEV1/FVC <0.7 and FEV1<50%)
* Severe renal disease (GFR < 15 ml/min)
* ejection fraction at baseline visit ≥ 50% by echocardiography or MRI
* Life expectancy < 1 year
* Pericardial disease
* Hypertrophic cardiomyopathy
* Myocardial infarction within the last 3 months
* Planned cardiac surgical intervention within 3 months after inclusion
* Geographical reasons (e. g. patients living outside Germany or planning to move abroad)
* Inability to give informed consent (e. g. mental disorders)
* Therapy with loop diuretics (e.g. torasemide, furosemide, piretanide) within 4 weeks prior to inclusion/baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The DZHK TransitionCHF Cohort Study will include patients with systolic dysfunction (NYHA I), i.e. (1) patients without a history of HF symptoms and (2) patients who reversed from symptomatic HF. Patients will be recruited prospectively at the participating DZHK centres, non-DZHK university hospitals and centers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of hospitalization for heart failure and cardiovascular death | 0.5 - 13 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Goettingen, Göttingen, Germany